CLINICAL TRIAL: NCT03428698
Title: Hyaluronic Acid and Amino Acid Gel Applied to the Alveolar Socket After Mandibular Third Molar Extraction Promotes Wound Healing: a Double Blind Randomized Controlled Clinical Trial
Brief Title: Hyaluronic Acid and Amino Acid Gel Applied to the Alveolar Socket After Mandibular Third Molar Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova, School of Dental Medicine (Other)
Responsible Party: Principal Investigator, Stefano Sivolella, DDS, PhD, MSc, University of Padova, School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1987/P
Record Dates: First submitted 2018-02-04; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Pain; Oral Surgery; Third Molar Extraction
Keywords: third molar extraction; hyaluronic acid
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental device (Experimental): The extraction was completed, the socket was filled with a topical amino acid + sodium hyaluronate gel (Aminogam®, sterile syringe 2 ml).
  Interventions: Device: Aminogam
- control no device (Placebo Comparator): The extraction was completed, socket was flushed, using a 2ml sterile syringe similar to one utilized to apply the gel, with sterile physiological solution.
  Interventions: Device: Aminogam

INTERVENTIONS:
Device: Aminogam — A lower third molar was extracted. All the surgical tools and materials as well as the surgical field were sterile. A full-thickness flap was raised and, if necessary, osteotomy and tooth sectioning were performed using a straight handpiece with dedicated burs under copious irrigation with sterile saline solution. The extraction was completed with curved and straight extractors, the socket was closely inspected and the dental follicle was removed. Depending on the group to which the patient was assigned, one of the following procedures was carried out.

SUMMARY:
Objective: The study aimed to assess the effect of topical application of an amino acid + sodium hyaluronate acid gel after lower third molar extraction.

Study design: 136 patients requiring lower third molar extraction were enrolled. An amino acid + sodium hyaluronate acid (HA) gel was applied to the sockets of the patients in the treatment group immediately following extraction; the sockets of the controls were simply flushed with a sterile saline solution. 7 and 14 days after surgery, patients' outcomes and postoperative complications were evaluated. Cumulative incidence of dehiscence and secondary outcome measures were analyzed using a chi-square test.

DETAILED DESCRIPTION:
A lower third molar was extracted under local anesthesia generally involving an inferior alveolar nerve block associated with a buccal nerve block (2% mepivacaine with 1:100,000 epinephrine, Optocain, Molteni Dental, Italy), plus sedation as necessary. All the surgical tools and materials as well as the surgical field were sterile. A full-thickness flap was raised and, if necessary, osteotomy and tooth sectioning were performed using a straight handpiece with dedicated burs under copious irrigation with sterile saline solution. The extraction was completed with curved and straight extractors, the socket was closely inspected and the dental follicle was removed. The bone edges were refined to remove the bone spurs with a bone lime and then irrigated with abundant sterile 0.9% saline solution. Depending on the group to which the patient was assigned, one of the following procedures was carried out: the socket was filled with a topical amino acid + sodium hyaluronate gel (Aminogam®, sterile syringe 2 ml) or the socket was flushed, using a 2ml sterile syringe similar to one utilized to apply the gel, with sterile physiological solution. The flap was then repositioned and sutured (Novosyn 4.0, B. Braun AG, Melsungen, Germany) to allow healing by primary intention. After surgery, the patients were prescribed antibiotics (amoxicillin clavulanate 1 g every 12 hours for 6 days, or clarithromycin 250 mg every 12 hours for 6 days) and painkillers (paracetamol 1000 mg every 8 hours was recommended). The patients were also provided standard postoperative recommendations regarding activity, diet, and smoking. The following data were registered at the time of surgery: the range of pre-operative mouth opening measurement (assessed by measuring the distance between the incisors), the type of sedation utilized, if osteotomy or root resection was carried out, the quantity of peri-operative bleeding, the amount of time between incision and suture (surgical procedure time).

ELIGIBILITY:
Inclusion Criteria:

* age 18 between 25 years,
* ASA I or II,
* necessitating lower wisdom tooth extraction,
* no evidence of inflammation

Exclusion Criteria:

* smoking more than 10 cigarettes a day,
* pregnancy,
* uncontrolled diabetes mellitus,
* any diseases contraindicating the surgical procedure,
* use of bisphosphonate,
* antibiotics or NSAIDs during the 30 days preceding surgery

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2009-09-10 (Actual); Primary Completion 2010-09-10 (Actual); Study Completion 2011-11-25 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of dehiscence | 14 days
  Surgical wound dehiscence is defined as a pathologic process consisting of a partial or complete disruption of the buccal and lingual mucosa layers of a surgical wound.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Sivolella, DDS, PhD, Principal Investigator — University of Padova
Locations (1):
- University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No